CLINICAL TRIAL: NCT04985799
Title: A Randomized Controlled Trial Comparing Retropubic KIM Sling to TVT Exact Midurethral Sling
Brief Title: Comparing KIM to TVT Exact Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-1324
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; Mixed urinary incontinence; Midurethral sling
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Gynecare TVT Exact sling (Active Comparator): Participants who are planning surgery for SUI are randomized to have placement of Gynecare TVT Exact sling and followed postoperatively for 1 year.
  Interventions: Device: Gynecare TVT Exact Continence System
- Neomedic KIM sling (Active Comparator): Participants who are planning surgery for SUI are randomized to have placement of retropubic Neomedic KIM sling and followed postoperatively for 1 year.
  Interventions: Device: Neomedic KIM (Knotless Incontinence Mesh)

INTERVENTIONS:
Device: Gynecare TVT Exact Continence System — Participants will have placement of Gynecare TVT Exact sling.
  Other Names: Midurethral sling
  Arms: Gynecare TVT Exact sling
Device: Neomedic KIM (Knotless Incontinence Mesh) — Participants will have placement of retropubic Neomedic KIM (Knotless Incontinence Mesh) sling
  Other Names: Midurethral sling
  Arms: Neomedic KIM sling

SUMMARY:
To assess to the non-inferiority of the retropubic Neomedic Knotless Incontinence Mesh (KIM) sling compared to the Gynecare Tension-free Vaginal Tape (TVT) Exact sling.

Participants: Women 21 years or older with a diagnosis of stress urinary incontinence (SUI) or mixed urinary incontinence (MUI) with objective evidence of SUI planning surgery for stress urinary incontinence.

Procedures (methods): Patients will be randomized to receive either the Gynecare TVT Exact sling or the retropubic Neomedic KIM sling. Patients will be followed for 1 year postoperatively.

DETAILED DESCRIPTION:
Midurethral slings (MUS) are recognized as a minimally invasive treatment of SUI. The retropubic route of MUS placement has a cure rate of 89.1% with long term subjective cure rates ranging from 51-88%. The Neomedic Knotless Incontinence Mesh (KIM) sling is a tension-free macroporous monofilament polypropylene knotless mesh designed to be resistant to elongation and deformation over time. The KIM sling also offers a reusable trocar, which results in less waste and cost- savings. KIM sling trocars are available for the retropubic route or trans-obturator (TOT) route.

While studies have been performed comparing the TOT approach of the KIM sling to other slings, no studies have been performed to date with the retropubic (RP) approach. The RP and TOT approaches to MUS have been shown to be equivalent in the treatment of SUI. Since the same mesh material of the KIM sling is used for both the TOT and RP approach, it can be hypothesis that the RP route would show similar treatment success rates.

A type 1 macroporous (> 75um) polypropylene mesh is the most appropriate material for vaginal implantation. However, literature has suggested that the design and weave of synthetic mesh material can also have a significant effect on efficacy and safety; therefore, the novel design of the KIM may be beneficial to reduce complications. If there is similar efficacy with the RP approach of the KIM sling to the TVT Exact, there will be benefit of reduced costs and the potential for less complications. With this study, the objective is to show non-inferiority of the KIM sling to the Gynecare TVT Exact.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than or equal to 21 years based on medical chart review
* Diagnosis of SUI or mixed urinary incontinence based on medical chart review
* Objective evidence of SUI as indicated by positive cough stress test or urodynamic stress incontinence during urodynamic testing within the last year prior to enrollment. Medical chart will be reviewed.
* Planning surgery for SUI with/without pelvic organ prolapse (POP) surgery

Exclusion Criteria:

* Current pregnancy, desire for future childbearing, less than or equal to 12 months postpartum at the time of enrollment
* Prior history of surgery for SUI based on medical chart review
* Bladder capacity <200 mL on Urodynamic testing or post-void residual (PVR) >150 mL on urodynamic testing or bladder scan.
* Non-ambulatory
* Current genitourinary fistula or urethral diverticulum based on pre-operative exam in the medical chart.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wu, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Christina Kunycky, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC Hospitals Hillsborough Campus, Hillsborough, North Carolina
  - Rex Hospital, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: Approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Padilla-Fernandez B, Garcia-Cenador MB, Gomez-Garcia A, Miron-Canelo JA, Gil-Vicente A, Silva-Abuin JM, Lorenzo-Gomez MF. Results of the surgical correction of urinary stress incontinence according to the type of transobturator tape utilized. Arch Ital Urol Androl. 2013 Sep 26;85(3):149-53. doi: 10.4081/aiua.2013.3.149. PMID 24085238
- [Background] Imamura M, Hudson J, Wallace SA, MacLennan G, Shimonovich M, Omar MI, Javanbakht M, Moloney E, Becker F, Ternent L, Montgomery I, Mackie P, Saraswat L, Monga A, Vale L, Craig D, Brazzelli M. Surgical interventions for women with stress urinary incontinence: systematic review and network meta-analysis of randomised controlled trials. BMJ. 2019 Jun 5;365:l1842. doi: 10.1136/bmj.l1842. PMID 31167796
- [Background] Ford AA, Rogerson L, Cody JD, Aluko P, Ogah JA. Mid-urethral sling operations for stress urinary incontinence in women. Cochrane Database Syst Rev. 2017 Jul 31;7(7):CD006375. doi: 10.1002/14651858.CD006375.pub4. PMID 28756647
- [Background] Richter HE, Albo ME, Zyczynski HM, Kenton K, Norton PA, Sirls LT, Kraus SR, Chai TC, Lemack GE, Dandreo KJ, Varner RE, Menefee S, Ghetti C, Brubaker L, Nygaard I, Khandwala S, Rozanski TA, Johnson H, Schaffer J, Stoddard AM, Holley RL, Nager CW, Moalli P, Mueller E, Arisco AM, Corton M, Tennstedt S, Chang TD, Gormley EA, Litman HJ; Urinary Incontinence Treatment Network. Retropubic versus transobturator midurethral slings for stress incontinence. N Engl J Med. 2010 Jun 3;362(22):2066-76. doi: 10.1056/NEJMoa0912658. Epub 2010 May 17. PMID 20479459
- [Background] Chapple CR, MacNeil S. The use of implanted materials for treating women with pelvic organ prolapse and stress urinary incontinence. Curr Opin Urol. 2019 Jul;29(4):431-436. doi: 10.1097/MOU.0000000000000619. PMID 30888974
- [Derived] Margulies SL, Osment AE, Bernard A, Schroeder MN, Askew AL, Agu IS, Kunycky CA, Geller EJ, Willis-Gray M, Chu CM, Wu JM. Noninferiority Randomized Clinical Trial: KIM Sling With Reusable Trocars Versus TVT Exact Sling. Urogynecology (Phila). 2025 Feb 1;31(2):101-107. doi: 10.1097/SPV.0000000000001596. Epub 2024 Nov 8. PMID 39514254

RESULTS

PARTICIPANT FLOW:
Groups:
- Gynecare Tension-free Vaginal Tape (TVT) Exact Sling: Participants who are planning surgery for stress urinary incontinence (SUI) are randomized to have placement of Gynecare Tension-free Vaginal Tape (TVT) Exact sling and followed postoperatively for 1 year.
  Gynecare TVT Exact Continence System: Participants will have placement of Gynecare TVT Exact sling.
- Neomedic Knotless Incontinence Mesh (KIM) Sling: Participants who are planning surgery for stress urinary incontinence (SUI) are randomized to have placement of retropubic Neomedic Knotless Incontinence Mesh (KIM) sling and followed postoperatively for 1 year.
  Neomedic KIM (Knotless Incontinence Mesh): Participants will have placement of retropubic Neomedic KIM (Knotless Incontinence Mesh) sling
Period: Overall Study
Arm/Group | Gynecare Tension-free Vaginal Tape (TVT) Exact Sling | Neomedic Knotless Incontinence Mesh (KIM) Sling
Started | 73 | 74
Completed | 73 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gynecare Tension-free Vaginal Tape (TVT) Exact Sling: Participants who are planning surgery for SUI are randomized to have placement of Gynecare TVT Exact sling and followed postoperatively for 1 year.
  Gynecare TVT Exact Continence System: Participants will have placement of Gynecare TVT Exact sling.
- Neomedic Knotless Incontinence Mesh (KIM) Sling: Participants who are planning surgery for SUI are randomized to have placement of retropubic Neomedic KIM sling and followed postoperatively for 1 year.
  Neomedic KIM (Knotless Incontinence Mesh): Participants will have placement of retropubic Neomedic KIM (Knotless Incontinence Mesh) sling
- Total: Total of all reporting groups
Arm/Group | Gynecare Tension-free Vaginal Tape (TVT) Exact Sling | Neomedic Knotless Incontinence Mesh (KIM) Sling | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (12.7) | 59.7 (12.1) | 58.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 74 | 147
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 63 | 62 | 125
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 74 | 147
Diabetes [Count of Participants; unit: Participants] | 6 | 8 | 14
Current smoker [Count of Participants; unit: Participants] | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success at 6 Weeks After Surgery
Description: Treatment success is defined by a composite outcome of 1) response of No or "no bother" to question #3 on urogenital distress inventory-6 (UDI-6) validated questionnaire AND no retreatment of stress incontinence.
Time Frame: 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecare Tension-free Vaginal Tape (TVT) Exact Sling | Neomedic Knotless Incontinence Mesh (KIM) Sling
Number analyzed (Participants) | 73 | 74
Participants | 61 | 51
Statistical Analysis 1: Comparison: Gynecare Tension-free Vaginal Tape (TVT) Exact Sling vs Neomedic Knotless Incontinence Mesh (KIM) Sling; Test type: Non-Inferiority — For the sample size, a total of 143 participants, or 72 participants per group was needed, based on a 90% effectiveness for both slings 14% non-inferiority margin, 80% power, alpha of 0.05 and a 20% dropout rate; p = 0.04, Chi-squared; Risk Difference (RD) = 14.8, 95% CI 2-sided [1.1 to 28.5]

2. Secondary Outcome: Number of Participants With Treatment Success at 1 Year After Surgery
Description: as for outcome 1
Time Frame: up to 1 year
Population: The overall number of participants analyzed was less than the number who completed the study at 6 weeks as some participants did not follow-up at 1 year. This outcome depended on completion of a questionnaire, which were collected on-line as well as during in-person visits. Thus, the number of participants analyzed for this secondary outcome was different than the number analyzed for the other secondary outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecare TVT Exact Sling | Neomedic KIM Sling
Number analyzed (Participants) | 67 | 71
Participants | 55 | 53
Statistical Analysis 1: Comparison: Gynecare TVT Exact Sling vs Neomedic KIM Sling; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.29, Chi-squared; Risk Difference (RD) = 7.4, 95% CI 2-sided [-6.2 to 21.1]

3. Secondary Outcome: Number of Participants Requiring Reoperation for Mesh Complications or Urinary Retention Thru 1 Year After Surgery
Description: Reoperation for mesh complications or urinary retention thru 1 year after initial sling surgery
Time Frame: up to 1 year
Population: The overall number of participants analyzed was less than the number who completed the study at 6 weeks as some participants did not follow-up at 1 year. This outcome measure was based on data collection from in-person visits, phone calls and electronic medical record review. Thus, the number of participants analyzed for this secondary outcome was different than the number analyzed for the other secondary outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecare TVT Exact Sling | Neomedic KIM Sling
Number analyzed (Participants) | 68 | 71
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Mesh Exposure Thru 1 Year After Surgery
Description: Sling mesh exposure identified on examination thru 1 year after surgery
Time Frame: up to 1 year after surgery
Population: The overall number of participants analyzed was less than the number who completed the study at 6 weeks as some participants did not follow-up at 1 year. Because this outcome measure required an in-person visit, the number of participants analyzed was lower than those for the other secondary outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecare TVT Exact Sling | Neomedic KIM Sling
Number analyzed (Participants) | 54 | 54
Participants | 6 | 1
Statistical Analysis 1: Comparison: Gynecare TVT Exact Sling vs Neomedic KIM Sling; Test type: Superiority; p = 0.11, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events are reported from after surgery until 1 year postoperative visit.
Description: Data collection occurred through 1 year after surgery for secondary outcomes and adverse events.
Arm/Group | Gynecare TVT Exact Sling | Neomedic KIM Sling
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/74
Other Adverse Events (participants affected / at risk) | 9/73 | 6/74
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gynecare TVT Exact Sling (N=73) | Neomedic KIM Sling (N=74)
Urinary retention (Renal and urinary disorders) | 3 (3) | 5 (5) — Voiding dysfunction after midurethral sling surgery
Mesh exposure (Renal and urinary disorders) | 6 (6) | 1 (1) — Vaginal mesh exposure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT04985799/Prot_SAP_000.pdf